CLINICAL TRIAL: NCT07313332
Title: Exploring Resistance Exercise Training Plus High-Intensity Interval Training (ReHIIT) as Cancer Prehabilitation: A Healthy Control Group Pilot Study
Brief Title: Exploring Resistance Exercise Training Plus High-Intensity Interval Training (ReHIIT) as Cancer Prehabilitation
Acronym: ReHIIT_CON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FMHS 237-0925
Record Dates: First submitted 2025-11-28; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy Adult Male and Female Volunteers; Intervention

STUDY DESIGN:
Intervention Model Description: Participants will complete 8-12 supervised sessions combining high-intensity interval cycling and resistance training (three sets of 8 reps @ ~70% 1-RM across 6 exercises (3 upper-body, 3 lower-body)).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance exercise training plus high-intensity interval training (ReHIIT) Intervention (Experimental): Participants will complete 8-12 supervised sessions combining high-intensity interval cycling and resistance training at 70% 1-RM.
  Interventions: Other: ReHIIT Training Intervention

INTERVENTIONS:
Other: ReHIIT Training Intervention — Participants will complete 8-12 supervised sessions combining high-intensity interval cycling (5 × 1-minute intervals at 110% CPET wattage, with 90-second rest intervals) and resistance training at 70% 1-RM (3 sets of 8-12 repetitions, 6 exercises).

SUMMARY:
Colorectal cancer is the fourth most common cancer in the UK. Prehabilitation, including exercise, can improve recovery from surgery. This pilot study investigates the combined effects of resistance and high-intensity interval training (ReHIIT) in healthy adults to establish baseline physiology and responses for comparison with cancer patients

DETAILED DESCRIPTION:
Colorectal cancers are a leading cause of death in the UK, but many can be cured with surgery alone. From diagnosis to surgery or alternative first treatment, the UK government mandates a maximum timeline of 31 days, providing only a short window in which patients may be physically optimised by exercise before surgery. There is increasing interest in clinical and academic settings regarding the potential benefits of exercise-based surgical prehabilitation. Although surgery is often successful, the combined effects of cancer and surgical stress can lead to poor clinical and patient-centred outcomes, including delayed return to normal activities and reduced quality of life. Physiological parameters known to be improved through exercise training, such as cardiorespiratory fitness and muscle mass, have been associated with more favourable clinical outcomes for individuals undergoing colorectal cancer surgery, including anaesthetic risk and tolerance to adjuvant treatment.

The limited time available before surgery remains a major challenge. Traditional modes of exercise training, including aerobic and resistance exercise performed separately, typically require six weeks or more to produce meaningful improvements in their primary physiological adaptations. As a result, recent cancer rehabilitation research has increasingly used high-intensity interval training (HIIT) because it requires less time and has been shown to improve both cardiorespiratory fitness and muscle mass more rapidly than traditional exercise modalities.

Although HIIT has demonstrated potential in several patient groups, previous work has shown that individuals with colorectal cancer may not experience improvements in cardiorespiratory fitness or muscle mass after a four-week HIIT intervention, even though the same protocol has produced adaptations in older adults and individuals with other cancer types. This may reflect a degree of anabolic or physiological resistance in the colorectal cancer population. Based on this, a current trial is comparing HIIT alone with a combined approach of HIIT plus resistance exercise training (ReHIIT) to determine whether the addition of resistance exercise can overcome this reduced adaptive response.

However, the expected magnitude of physiological adaptation to four weeks of ReHIIT in adults without cancer has not been fully characterised. This study will therefore explore changes in cardiorespiratory fitness, muscle mass, and associated metabolic and molecular mechanisms in healthy adults following a four-week ReHIIT programme.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Availability and willingness to attend the Royal Derby Hospital site for a minimum of 8 exercise sessions and 2 assessment sessions across the study period.

Exclusion Criteria:

* BMI <18 or >35 kg/m2
* Known active cance
* Known metabolic disease
* Current known neurological or musculoskeletal conditions (e.g. epilepsy)
* Active known cardiovascular, cerebrovascular or respiratory disease - e.g:
* Uncontrolled hypertension (systolic BP > 160 mmHg or diastolic BP >100 mmhg)
* Myocardial infarction within the last 6 months or unstable angina
* Heart failure (New York Heart association Class III/IV)
* Arrhythmia
* Right to left cardiac shunt
* Aneurysm of a named blood vessel
* COPD
* Pulmonary hypertension
* Exercise-induced or brittle asthma
* Previous stroke/transient ischaemic attack
* Abnormal ECG results (at the discrepancy of the study doctor)
* Patients who are unable to undergo CPET based on ATS/ACSS guidelines ^
* Pre-existing clotting disorder known to the participant or anticoagulant use
* Family history of severe bleeding requiring medical intervention
* Participation in a research study in the last 3 months involving invasive procedures or an inconvenience allowance (ALL UoN FMHS UREC approved studies)
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in anaerobic threshold (CPET-derived) | From baseline to 4-weeks after the start of the intervention
Change in Muscle mass | From baseline to 4-weeks after the start of the intervention
  Derived from DXA and stable isotope assessments of muscle mass (COSIAM, Cegielski et al., 2021)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Bethan E Phillips, Principal Investigator — University of Nottingham
Locations (1):
- Medical School, University of Nottingham, Royal Derby Hospital, Derby, Derbyshire, United Kingdom